CLINICAL TRIAL: NCT05712226
Title: Single-center Evaluation of Sleepiz One+ in Measuring Respiration Rate and Heart Rate Compared to Gold Standard
Brief Title: Sleepiz One+ Versus Capnography and Electrocardiography
Acronym: SPZCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sleepiz AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22-007-CI
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: COPD; Hypertension; Sleep Apnea; Asthma; Heart Diseases; Respiratory Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension; Sleep Apnea Syndromes; Asthma; Heart Diseases; Respiration Disorders

STUDY DESIGN:
Masking Description: Annotators of capnography data were blinded to the values provided by the investigational device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleepiz One+ vs. gold standard (Other): Each enrolled participant will undergo a simultaneous recording with the Sleepiz One+, Capnography device and cardiorespiratory polygraphy with reduced number of channels (ECG and REB only) to measure respiration rate at and heart rate at rest, while sitting and lying down on a bed.
  Interventions: Device: Sleepiz One+

INTERVENTIONS:
Device: Sleepiz One+ — In this study Sleepiz One+ will measure heart rate and respiration rate of a participant sitting or lying in different positions (right and left side, back, abdomen) on a bed. The recording will take around 35 minutes.

SUMMARY:
EtCO2, or exhaled carbon dioxide, is a non-invasive and commonly used measure for respiratory rate and function. It can be easily monitored using a device called a capnograph, which consists of a sensor that is placed near the patient's mouth or nose and a monitor that displays the concentration of carbon dioxide in the respiratory gases in real-time.

EtCO2 capnography is generally considered a reliable and accurate method for monitoring respiration and is often used as a gold standard for comparing the performance of other methods for measuring respiration.

Therefore, the primary aim of this study is to provide a thorough comparison of the performance of Sleepiz One+ and EtCO2 Capnography for measuring respiration rate, in healthy adults and patients suffering from chronic conditions (e.g. hypertension, COPD, asthma, diabetes), at rest in a clinical setting. Additionally, the performance of heart rate estimation will be evaluated against ECG.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Age >=18years
* Informed Consent as documented by signature
* One (or more) chronic medical condition/s (e.g., diabetes, asthma, cardiovascular or respiratory diseases, etc.)

Healthy volunteers

* Age >=18years
* Informed Consent as documented by signature
* No diagnosed chronic medical condition

Exclusion Criteria:

Patients

* Previous enrolment into the current study,
* Cardiac pacemaker or another implanted electrical device
* Women who are pregnant or breastfeeding
* Inability to follow the procedures of the study, e.g., due to language problems, psychological disorders, dementia, delirium etc. of the participant

Healthy volunteers:

* Previous enrolment into the current study,
* Cardiac pacemaker or another implanted electrical device
* Women who are pregnant or breastfeeding
* Inability to follow the procedures of the study, e.g., due to language problems, psychological disorders, dementia, delirium etc. of the participant
* Presence of diagnosed chronic medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Respiration rate measurement accuracy per 60s epoch against visually scored capnography data, recorded on subjects lying down and resting on a bed. | 60s

CONTACTS AND LOCATIONS:
Locations (1):
- Schlaflabor Fluntern, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No